CLINICAL TRIAL: NCT03139513
Title: Survival in Adult Patients With BRAF V600 Mutation-Positive Advanced Melanoma: A Non-Interventional Ambispective Study of a Cohort of Patients Treated With Cobimetinib During the French Early Access Program (TAU)
Brief Title: A Study of Adult Participants With BRAF V600 Mutation-Positive Advanced Melanoma Treated With Cobimetinib (Cotellic®) During the French Early Access Program (Temporary Authorization for Use [TAU])
Acronym: MELANIS
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29964
Record Dates: First submitted 2017-05-02; First posted 2017-05-04 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — cobimetinib; Vemurafenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Metastatic Melanoma: Participants with BRAF V600 mutation-positive unresectable or metastatic melanoma, having started treatment with cobimetinib in combination with vemurafenib as per local guidelines and/or routine clinical practice in context of TAU program, will be observed.
  Interventions: Drug: Cobimetinib; Drug: Vemurafenib

INTERVENTIONS:
Drug: Cobimetinib — Participants will receive cobimetinib as per local guidelines and/or routine clinical practice.
  Other Names: Cotellic®
Drug: Vemurafenib — Participants will receive vemurafenib as per local guidelines and/or routine clinical practice.
  Other Names: Zelboraf®

SUMMARY:
This is a multicentre, ambispective (both retrospective and prospective), and non-interventional study conducted in France in adult participants with BRAF V600 mutation-positive unresectable or metastatic melanoma treated with cobimetinib in combination with vemurafenib (Zelboraf®).

DETAILED DESCRIPTION:
Concomitantly to the marketing authorization applications for cobimetinib and vemurafenib to European Medicines Agency (EMA) and United States Food and Drug Administration (USFDA) in 2014, a French TAU program was initiated in February 2015. This study will enroll participants under this program.

ELIGIBILITY:
Inclusion Criteria:

* Participants included in the TAU from 26 February 2015
* Participants with BRAF V600 mutation-positive unresectable or metastatic melanoma treated with cobimetinib in combination with vemurafenib
* For alive participants: participants who have been informed verbally and in writing about this study who do not object to their data being electronically processed or subjected to data quality control
* For participants who died before the inclusion period: participants who did not express their opposition when they were alive

Exclusion Criteria:

- Alive participants unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with BRAF V600 mutation-positive advanced melanoma treated with cobimetinib during the French early access program (TAU).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-10-27 (Actual); Primary Completion 2018-08-22 (Actual); Study Completion 2018-08-22 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | From first intake of cobimetinib up to date of death due from any cause (assessed up to 18 months)

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors (RECIST) | From first intake of cobimetinib up to first disease progression or death from any cause (assessed up to 18 months)
Percentage of Participants with Complete Response (CR) or Partial Response (PR) to Treatment According to RECIST as Assessed by Physician | From first intake of cobimetinib up to first disease progression or death from any cause (assessed up to 18 months)
Time to Cobimetinib Treatment Discontinuation | From first intake of cobimetinib up to cobimetinib treatment discontinuation (assessed up to 18 months)
Percentage of Participants by Treatments After Disease Progression or Permanent Cobimetinib Treatment Discontinuation | From disease progression or permanent cobimetinib treatment discontinuation up to overall study completion (assessed up to 18 months)
Retrospective Period: Percentage of Participants with Targeted Adverse Events (AEs) | From first intake of cobimetinib up to inclusion in the study (up to Day 1)
  An AE is defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Participants with following targeted adverse events will be reported: fever (pyrexia), diarrhea, hepatic abnormalities, creatinine phosphokinapse (CPK) increased, rhabdomyolysis, retinal serous detachment, decrease in left ventricular ejection fraction (LVEF), squamous cell skin carcinoma and keratoacanthom, renal failure, drug reaction (or rash) with eosinophilia and systemic syndrome (DRESS), rash not otherwise specified (NOS), and photosensitivity.
Prospective Period: Percentage of Participants with Adverse Events (AEs) | From first intake of cobimetinib up to overall study completion (assessed up to 18 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (33):
- France (33):
  - Centre Hospitalier d'Albi, Albi
  - Hopital Prive D Antony; Dermatologie, Antony
  - Chic Cote Basque Bayonne; Medecine II, Bayonne
  - CHU Besançon - Hôpital Jean Minjoz, Besançon
  - Hopital Avicenne; Dermatologie, Bobigny
  - CH Fleyriat, Bourg-en-Bresse
  - CH Metropole de Savoie, Chambéry
  - Chu Estaing; Dermatologie, Clermont-Ferrand
  - Hopital Louis Pasteur; Sce Dermatologie, Colmar
  - Centre Georges Francois Leclerc, Dijon
  - Chu Site Du Bocage;Dermatologie, Dijon
  - Centre Hospitalier Le Mans; Dermatologie, Le Mans
  - Hopital Claude Huriez; Sce Dermatologie, Lille
  - CHU de Limoges - Hôpital Dupuytren, Limoges
  - Hopital Timone Adultes; Dermatologie, Marseille
  - Hopital Jacques Monod; Dermatologie, Montivilliers
  - Hopital Saint Eloi; CHU de Montpellier; Svc de Dermatologie, Montpellier
  - CH de Mulhouse Hôpital Emile Muller, Mulhouse
  - Hopital l Archet 2; Ginestriere, Service de; Dermatologie, Nice
  - Hopital Cochin; Dermatologie, Paris
  - Groupe Hospitalier Bichat Claude Bernard, Paris
  - CENTRE HOSPITALIER ANNECY-GENEVOIS; Dematologie, Pringy
  - Centre Eugene Marquis Centre Regional de Lutte Contre Le Cancer, Rennes
  - CHU Rouen - CH C. Nicolle - Clinique dermatologique, Rouen
  - CHU de Saint-Etienne - Hopital Nord, Saint-Etienne
  - CHI de Poissy St Germain, Saint-Germain
  - Hopital Broussais, St-Malo
  - Pole de Cancerologie Prive Strasbourgeois, Strasbourg
  - Hopital Bel Air, Thionville
  - Hia Sainte Anne; Medecine Interne Oncologie, Toulon
  - CHU de Toulouse - Hôpital Larrey, Toulouse
  - Centre Hospitalier Valence, Valence
  - Institut Gustave Roussy; Dermatologie, Villejuif